CLINICAL TRIAL: NCT07225270
Title: A Randomized, Open-Label, Phase 3 Study of Rinatabart Sesutecan (Rina-S) Plus Standard of Care Versus Standard of Care as Maintenance Treatment After 2L Platinum-Based Doublet Chemotherapy in Participants With Recurrent Platinum-Sensitive Ovarian Cancer (PSOC)
Brief Title: Study to Assess the Efficacy and Safety of Rina-S Plus Standard of Care Compared to Standard of Care for Maintenance Treatment of Participants With Recurrent Platinum-sensitive Ovarian Cancer After Second-line (2L) Platinum-based Doublet Chemotherapy
Acronym: RAINFOL-04
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCT1184-04; 2025-522167-15-00 (EU CTIS Number); jRCT2051250197 (Registry Identifier: Japan Registry for Clinical Trials (jRCT)); GOG-3134 (Other: Other Sponsor Identifier); ENGOT-OV96 (Other: Other Sponsor Identifier)
Record Dates: First submitted 2025-11-04; First posted 2025-11-06 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Cancer; Platinum-sensitive Ovarian Cancer; PSOC
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rina-S + SOC (Experimental): Participants will receive Rina-S and SOC consisting of either bevacizumab maintenance or no maintenance treatment (observation).
  Interventions: Drug: Rina-S; Drug: Bevacizumab
- SOC (Active Comparator): Participants will receive SOC consisting of either bevacizumab maintenance or no maintenance treatment (observation).
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Rina-S — Intravenous (IV) infusion
  Other Names: Rinatabart sesutecan; GEN1184; PRO1184
  Arms: Rina-S + SOC
Drug: Bevacizumab — IV infusion

SUMMARY:
This Phase 3 study will be conducted in different countries around the world with up to about 528 participants.

The purpose of this study is to evaluate how well Rina-S works against ovarian cancer in combination with available standard of care therapy that is already approved and used for ovarian cancer.

Participants will receive either Rina-S monotherapy (by itself), Rina-S plus bevacizumab, bevacizumab (standard of care) by itself, or no treatment (only monitoring, also standard of care). No participants will be given placebo. Participants will participate in 1 of 2 arms.

The treatment duration will be different for every participant. If a participant's cancer stays the same or gets better, and there are not any serious problems, participants can keep getting study treatment for as long as the study is open.

Participants will be asked to attend 1 to 3 visits at the study clinic for each cycle (duration of cycle is 3 weeks). During visits, there will be various tests (such as blood draws) and procedures (such as recording of heart activity and imaging) to monitor whether the study treatment is safe and effective. The overall study duration (including screening, treatment, and follow-up) for each participant will be different for every participant.

DETAILED DESCRIPTION:
This is a randomized, open-label, Phase 3 study of Rina-S + standard of care (SOC) versus SOC as maintenance treatment after second-line (2L) platinum-based doublet chemotherapy in participants with recurrent PSOC.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have histologically or cytologically confirmed high-grade serous or endometrioid epithelial ovarian cancer (EOC), primary peritoneal cancer, or fallopian tube cancer.
* Must have PSOC defined as progressive disease > 6 months (ie, 183 days) from the last dose of primary (first-line [1L]) platinum therapy.
* Participants with known breast cancer (BRCA)-mutated (somatic or germline) or homologous recombination deficiency (HRD)-positive ovarian cancer who achieved complete response (CR)/no clinical evidence of disease (NED) or partial response (PR) following 1L platinum-based chemotherapy regimen must have previously received PARPi maintenance therapy as part of their 1 L treatment.
* Must have completed platinum-based chemotherapy in the 2L treatment for recurrent PSOC.
* Must have received platinum-based chemotherapy in the 1L treatment and received platinum-based chemotherapy in the 2L treatment.
* Must be randomized no later than 8 weeks from the last dose of the 2L platinum-based therapy.
* Participants must have achieved a CR/NED, PR, or SD, as assessed by the investigator, following completion of 2L platinum-based chemotherapy.

Key Exclusion Criteria:

* Participants with clear cell, mucinous, or sarcomatous histology, mixed tumors containing any of the above histologies, or low-grade/borderline ovarian tumors
* More than 2 prior lines of systemic therapy.
* Progression while on or following 2L platinum-based regimen prior to randomization.
* Participants who receive an intervening systemic anticancer treatment (excluding bevacizumab) after the last dose of 2L platinum-based chemotherapy and prior to randomization.

Note: Other protocol-defined Inclusion and Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2026-03-16 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1, as Determined by Investigator Assessment | Up to approximately 3 years

SECONDARY OUTCOMES:
Overall Survival | Up to approximately 4 years
PFS, per RECIST 1.1, as Determined by Blinded Independent Central Review | Up to approximately 3 years
Second Determination of PFS (PFS2) | Up to approximately 4 years
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to approximately 4 years
Overall Change from Baseline in Global Health Status (GHS)/Quality of Life (QoL) Score Using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) Questionnaire | Up to approximately 4 years
Time to Deterioration (TTD) in the GHS/QoL Score Using the Quality of Life Questionnaire Core 30 Questionnaire | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (2):
- Mt. Sinai Comprehensive Cancer Center, Miami, Florida, United States
- Osaka Medical and Pharmaceutical University Hospital, Takatsuki, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No